CLINICAL TRIAL: NCT05245253
Title: The Immune Response of the Human Brain in Survivors of Critical Illness
Brief Title: Trauma and Critical Care Exposure Examined With PET (TRAPETS)
Acronym: TRAPETS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jessica Kåhlin, Principal Investigator, Attending in ICU, Karolinska University Hospital
Other Study IDs: 2019-04228
Record Dates: First submitted 2021-02-17; First posted 2022-02-17 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Cognitive Dysfunction; Critical Illness; Trauma
MeSH Terms: conditions — Cognitive Dysfunction; Critical Illness; Wounds and Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood from subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients: Trauma patients 20-60 years of age
  Interventions: Radiation: Positron Emission tomography

INTERVENTIONS:
Radiation: Positron Emission tomography — Patients will be tested with PET-examination at 3 weeks, 3 months and 1 year after the trauma

SUMMARY:
The overall aim is to examine the impact of trauma and critical illness on the brain, peripheral immune system and cognition. This is a prospective study where a study group exposed to trauma and intensive care will be be examined with consecutive PET imaging, EEG, biomarkers and cognitive testing within 3 weeks of the trauma, after 3 months and finally after 12 months. The study group will consist of twenty trauma patients treated in the intensive care unit.

DETAILED DESCRIPTION:
Background Cognitive impairment is a common problem after an episode of critical illness. Cognitive impairment occurs regardless of diagnosis of admission and this profound impairment is comparable to a traumatic brain injury or Alzheimers disease. For specific diagnoses, such as sepsis and ARDS, long-term cognitive dysfunction occurs in 50-70% of patients. Exposure to trauma without traumatic brain injury results in long-term cognitive impairment in every second patient and seemingly regardless of trauma severity.

The cognitive impairment persists for >6 months in 36% and >12 months in 25% of patients, demonstrating a long-term effect of critical illness.

Multiple domains of cognitive dysfunction are involved but the pattern of brain injury is not fully described. Neuroimaging with magnetic resonance imaging show cortical and subcortical lesions, generalized and focal atrophy in hippocampus and superior frontal lobes along with spread white matter lesions.

Underlying mechanisms of brain injury in ICU-survivors without head trauma or stroke but with cognitive impairment are hypoxia, hypoglycemia, hypothermia and/or inflammation. Peripheral injury and inflammation causes neuronal injury by release of cytokines and by inducing programmed cell-death in hippocampus , a region essential for memory and also demonstrated to be particularly sensitive to damage during endotoxemia.

Sterile injury such as surgery affects the central nervous system by disruption of blood-brain barrier integrity and further invasion of macrophages. The signaling from periphery to brain with cytokines induces microglia activation, detectable with positron emission tomography (PET) using ligands targeting the translocator protein (TSPO). Using this method it was demonstrated that surgical patients had a downregulation of glia activation in the early postoperative period and a subsequent upregulation of the brain immune system 3 months postoperatively . This upregulation was also linked to certain domains of cognitive dysfunction.

The impact of critical illness on the brain immune system is poorly understood. In critical illness and trauma, there is substantial release of chemokines and cytokines that affect the immune system and subsequently the brain and cognitive functions.

Rationale of study Previous findings in animals and in the human brain post-surgery demonstrate that immune cells in the brain are activated by a sterile peripheral injury, shown with PET imaging techniques. Animal studies indicate that neuroinflammation and local intracranial cytokine release occur after critical illness. However, this is not investigated in humans after critical illness. Furthermore, no data is available on the connection between neuroinflammation and cognitive dysfunction after critical illness. This study is therefore outlined to study the human brain and its immune cell activation after critical illness using PET imaging. Further, this study aims at mapping the trajectory of systemic inflammatory mediators, markers of neurodegeneration and brain injury and correlate this with cognitive dysfunction after critical illness.

Because ICU survivors frequently display long-term cognitive decline affecting quality of life, there is a need to understand the impact of unresolved brain immune activation on cognitive outcome. As the probability to survive severe trauma and critical illness increases, this group of patients enlarges, proposing an increased challenge on health care, rehabilitation and society. Notably, this project is the first to translate results from animal ICU models of brain immune activation and local intracranial cytokine release to the human ICU population. The investigators hope to provide novel insights and a more comprehensive understanding of the link between human brain immune activation, peripheral immune activation and cognitive dysfunction after trauma and critical illness.

Hypothesis The investigators hypothesize that unresolved brain immune activation in trauma patients after intensive care treatment closely associates with persistent cognitive decline.

Objectives and purposes The overall aim is to examine the impact of trauma and critical illness on the brain, peripheral immune system and cognition.

The specific aims are:

1. To examine the trajectory of trauma-induced neuroinflammation and subsequent long-term cognitive decline in ICU-survivors.
2. To explore the relationship between acute systemic inflammatory biomarker patterns and later neuroinflammation with long-term cognitive decline.
3. On the basis of 1 and 2, identify systemic inflammatory reaction patterns that associate with unresolved neuroinflammation and cognitive decline 12 months after trauma.

Detailed objectives The objective is to study cerebral immune cell activation using the cell specific PBR probe detected with PET imaging techniques.

Selected key areas of the brain involved in short term memory, attention and executing functions will be targeted, being the most affected in cognitive dysfunction after critical illness.

These findings will be correlated with cognitive dysfunction in ICU-survivors and with systemic inflammatory biomarkers present in blood.

Study design Type and design of the study This is a prospective study where a study group exposed to trauma and intensive care will be be examined with consecutive PET imaging and biomarkers and cognitive testing within 3 weeks of the trauma, after 3 months and finally after 12 months. The study group will consist of twenty trauma patients treated in the ICU.

General study outline and study schedule Twenty adult (20-60 years) male and female trauma patients with an ISS-score of more than 15, admitted to an intensive care unit will be included. A member of the research group will recruit the patients on dismissal from the ICU or after arrival on the ward after an interview. Upon inclusion, data and blood samples from the admission in the trauma room and on the ICU will be collected. PET-exams will be performed after 14 days post trauma, after 3 months and after 1 year. Cognitive testing will also be performed on these occasions, as well as blood sampling.

Patients 20-60 years old with an ISS-score of Inclusion criteria of ≥15 and treated in the ICU for >24h will be asked for informed consent. Exclusion criteria are traumatic brain injury, neuropsychiatric disorder, previous stroke, severe comorbidities, terminal malignancy, high dose steroid treatment or presumed uncooperativeness or legal incapacity.

Subject withdrawal Study subjects are free to permanently discontinue their participation in the scheduled study assessments at any time without providing a reason. Their legal representatives can permanently discontinue the study subjects as well. The study subjects can also permanently discontinue their participation in the study if the investigator recommends it for any medical reason.

Detailed Study Description After inclusion, a physician in the research group will place a note in the medical record (Take Care, i.e. Karolinska University Hospital Medical Record System) describing that the patient has been included in the current study. All following parts of the study protocol, vital sign data, cognitive test results, laboratory tests and related information on organ system functions, pain, medication and sleep will be recorded in an electronic CRF and kept on a computer for further analysis.

All trauma patients with a severe trauma will arrive in the Trauma Unit at the Trauma Center at Karolinska University Hospital, Solna, Stockholm and will undergo routine assessment and acute trauma care management according to ATLS (Advance Trauma Life Support)-guidelines. Screening blood samples are drawn from all patients after arrival in the Trauma Unit. After a primary and secondary survey a CT will be performed unless urgent surgery is performed in advance. Subsequently the patient is referred to the ICU. On admission, screening blood samples are drawn and scores of organ dysfunction are registered. After inclusion (at discharge from the ICU or at the ward) data and blood samples from the admission in the trauma room and on the ICU will be collected.

On inclusion, detailed parameters on previous illnesses, ICU-parameters and prescribed medications will be registered.

On inclusion a blood sample will be drawn and sent for genetic analysis of polymorphism of the translocator protein (TSPO), which is the target of the radio ligand used at the PET-exaxminations. This protein has different expressions with different affinity for the (11C) PBR28 radio ligand, affecting the signal of the PET-examination. Low-affinity binders will be excluded from the trial.

The patient will thereafter be scheduled for the first PET scanning (≤1month after the trauma), which includes an initial MRI scan and formation of an individual helmet for the PET scan procedure. After arriving in at the PET unit the following is performed:

1. A cognitive test (according to the CANTAB protocol) 2. Routine vital signs are recorded as well as body weight, length and BMI. 3. Arterial or venous blood sampling (a total volume of 20 mL whole blood for inflammatory biomarkers, ex vivo tests of inflammatory reactivity and additional 10 mL for genetic analysis of inflammatory biomarkers

1. PET-imaging: PET-examinations will be performed at 3 weeks, 3 months and 12 months. We will use the (11C) PBR28 radio ligand that targets (TSPO), leading to information on glia activation in specific regions of the brain. The ligand is injected intravenously and blood is sampled through and arterial cannula for determination of peripheral levels of the ligand. The first PET-examination is preceded by an MRI scan for co-registration with PET and definition of anatomical regions. The patient will be positioned in the PET-system using an individual helmet that allows for no head movements during the procedure.

   During image processing, regions of interest (ROIs) will be defined. Brain areas of interest for cognitive function will further be assessed, such as hippocampus, lateral frontal cortex, lateral parietal cortex and putamen.
2. Cognitive testing: The Cambridge Neuropsychological Test Automated Battery (CANTAB) will be used to determine cognitive dysfunction in various modalities, such as general memory and learning, working memory and executing function, visual memory, attention and reaction time, verbal memory and decision making. The test battery is computer-based and validated and a standard method in cognitive testing.
3. Systemic inflammatory biomarkers: Blood sampling will take place on arrival to the trauma unit, daily at the ICU at 21 days and at 3 months and 12 months. Blood borne immune cells will be collected for later analysis of immune cell phenotypes (e.g. M1-M2 transition and T-regulatory cell populations). Inflammatory molecules will be mapped (CRP, pro-calcitonin, LPK, IL-1, IL-6, IL-10, HMGB1, TNFa) and furthermore markers of neurodegeneration (b-amyloid, tau), markers of brain injury (e.g. S100, GFAP, NSE, NFL, UCH-L1, BDNF) and biochemical markers for kidney function, liver function and coagulation.

Data analysis: The percentage change in distribution volume (VT) for the (11C) PBR28-ligand between the three time points will be analyzed with repeated measures analysis of variance. Post-hoc tests for individual ROIs will be performed using paired t-tests. The percentage change of VT will be related to corresponding changes in cognitive test variables using Pearson correlation analysis. A similar correlation between changes in VT and blood biomarkers of inflammation will be performed with Pearson correlation analysis.

Principal component analysis will be used to reduce the dimensionality of biomarker data and to gain insight into the correlation between neuroinflammation and cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 20-60 years of age.
2. Trauma with an ISS score of ≥15
3. Informed consent

Exclusion Criteria:

1. Patient´s refusal to participate in the trial
2. Any traumatic brain or spinal injury prior to admission
3. Disabling neuropsychiatric disorder (dementia-diagnosis, Mb Alzheimer, Mb Parkinson, schizophrenia or severe mental depression prior to ICU admission)
4. Any preadmission history of stroke with neurological sequelae
5. Co-morbidities prior to ICU admission such as severe cardiac, hepatic, hematological or renal impairment
6. Terminal phase of chronic disease or malignancy
7. High-dose steroid treatment before ICU admission or during ICU care
8. Presumed uncooperativeness or legal incapacity

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Trauma patients in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Neuroinflammation | 3 weeks-12 months post trauma
  The trajectory of neuroinflammation as measured by repeated PET-examinations. More specifically, the probe targeting the translocator protein indicates microglia-activation as a sign of inflammatory activation. The change in binding capacity of the probe will be measured, generating a difference in signal in the regions of interest.
Cognitive dysfunction | 3 weeks-12 months post trauma
  Cognitive function will be evaluated with Cambridge Neuropsychological Automated Battery (CANTAB) with five different tests at three timepoints. A z-score will be calcualted for each test and then aggregated into a total z-score for the entire test.

CONTACTS AND LOCATIONS:
Overall Officials: Lars I Eriksson, Professor, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Perioperative Medicine and Intensive Care, Stockholm, Sweden

REFERENCES:
- [Result] Forsberg A, Cervenka S, Jonsson Fagerlund M, Rasmussen LS, Zetterberg H, Erlandsson Harris H, Stridh P, Christensson E, Granstrom A, Schening A, Dymmel K, Knave N, Terrando N, Maze M, Borg J, Varrone A, Halldin C, Blennow K, Farde L, Eriksson LI. The immune response of the human brain to abdominal surgery. Ann Neurol. 2017 Apr;81(4):572-582. doi: 10.1002/ana.24909. Epub 2017 Apr 11. PMID 28253549
- [Result] Owen DR, Yeo AJ, Gunn RN, Song K, Wadsworth G, Lewis A, Rhodes C, Pulford DJ, Bennacef I, Parker CA, StJean PL, Cardon LR, Mooser VE, Matthews PM, Rabiner EA, Rubio JP. An 18-kDa translocator protein (TSPO) polymorphism explains differences in binding affinity of the PET radioligand PBR28. J Cereb Blood Flow Metab. 2012 Jan;32(1):1-5. doi: 10.1038/jcbfm.2011.147. Epub 2011 Oct 19. PMID 22008728